CLINICAL TRIAL: NCT04444492
Title: Long-term Need of Ranibizumab Injections With or Without Early Targeted Peripheral Laser Photocoagulation for Treatment of Macular Edema Due to Central Retinal Vein Occlusion
Brief Title: Combination of Ranibizumab and Targeted Laser Photocoagulation
Acronym: CoRaLaII
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CoRaLaII
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Central Retinal Vein Occlusion With Macular Edema
Keywords: retinal vein occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinded BCVA assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab+Laser-arm (Experimental): Ranibizumab injections and additional targeted laser
  Interventions: Drug: Ranibizumab Injection; Device: Laser photocoagulation
- Ranibizumab-arm (Active Comparator): Only Ranibizumab injections
  Interventions: Drug: Ranibizumab Injection

INTERVENTIONS:
Drug: Ranibizumab Injection — initial three injections of Ranibizumab - afterwards pro re nata monthly
  Other Names: Lucentis
Device: Laser photocoagulation — Areas of capillary non-perfusion will be treated with photocoagulation upto 4 times
  Arms: Ranibizumab+Laser-arm

SUMMARY:
Intravitreal injections of Ranibizumab will be applied in all patients according to treatment guidelines. The experimental group will receive additional targeted laser photocoagulation of the peripheral areas of capillary non-perfusion (up to 4 laser treatments within 1st year of the study). Based on the long-term observation after CoRaLa I study an importantly shorter duration of treatment and a relevant reduction of the total number of re-injections in RL patients is expected.

DETAILED DESCRIPTION:
Retinal vein occlusion (RVO) is the second most common retinal vascular disease leading to visual impairment. Main cause for visual impairment in CRVO (Central Retinal Vein Occlusion) is macular edema (ME) while neovascularization of the retina and/or the anterior segment is the most serious complication leading to vitreous hemorrhage, retinal detachment and neovascular glaucoma. In serious cases loss of vision is imminent. To date, no causal treatment has been proven to be effective in large trials. Intravitreal injections of drugs that inhibit the vascular endothelial growth factor (VEGF) and other inflammatory factors are the current treatments of choice for ME due to CRVO. Two different anti-VEGF drugs (ranibizumab and aflibercept), and a biodegradable dexamethasone implant are approved by the EMA (European Medicines Agency). Based on data from confirmatory studies anti-VEGF-drugs are recommended as a treatment of first choice in patients with RVO. All intravitreal drugs provide only a temporary effect with need for re-treatment for recurrences of ME. Mean number of ranibizumab application needed in CRVO patients was found to be 7.4 to 10.2 injections in 12 months. A significant number of CRVO patients require treatment over several years. Need for repetitive treatments and ophthalmic controls are a major burden for patients (and their relatives who are required for driving the patients to ophthalmologists) despite of only few adverse events and generally well-tolerated injections. Endophthalmitis is the most severe ocular complication which can be eye-sight-threatening. The more injections are administered, the higher is the cumulative risk of complications. Due to high costs (>1000 € per injection) treatment with repeated injections over years is of significant socio-economic importance, too. Therefore, treatments concepts which would lead to permanent reduction of ME and/or significantly reduce the number of re-injections over long-term periods are the major currently unmet need in patients with RVO.

Until now, several studies evaluated the impact of the additional pan-retinal laser photocoagulation in patients undergoing the anti-VEGF-treatment for the ME due to retinal vein occlusions. However, most of the studies are limited by retrospective design, small number of evaluated patients or lack of the randomization. None of the available prospective randomized studies had sufficient power to finally clarify the benefit of the additional laser treatment. Therefore, there is an unmet need for a large randomized, prospective, multicentric trials.

The proposed study will be the first sufficiently powered trial evaluating the long-term effect of targeted laser photocoagulation performed selectively (targeted) in peripheral areas of non-perfusion in combination with standard anti-VEGF treatment (ranibizumab injections) on the duration of the required intravitreal treatment over time period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of macular edema due to central retinal vein occlusion foveal thickness > 250 μm (measured by OCT)
* Age > 18 years
* Written informed consent of the patient
* BCVA score in the study eye between 24 letters (20/320) and 78 letters (20/25) measured in ETDRS chart
* History of CRVO no longer than 6 months
* Presence of capillary non-perfusion in peripheral retina larger than 5 disc areas documented in ultra wide-field fluorescein angiography
* Ability and willingness to attend all scheduled visits and assessments

Exclusion Criteria:

* CRVO with ischemic maculopathy defined as diameter of the foveolar avascular zone larger than 2 optic disc diameters
* Macular edema due to another etiology than retinal vein occlusion (e.g. diabetic maculopathy, uveitis, age related macular degeneration, Irvine-Gass syndrome)
* History of idiopathic central serous chorioretinopathy
* Presence of vitreoretinal interface disease (e.g. vitreomacular traction, epiretinal membrane), either on clinical examination or in OCT
* An eye that, in the investigator's opinion, would not benefit from resolution of macular edema, such as eyes with foveal atrophy, dense pigmentary changes, or dense subfoveal hard exudates
* Aphakia in the study eye
* Scatter laser photocoagulation or macular photocoagulation in the study eye prior to study entry
* Intraocular or periocular injection of steroids in the study eye prior to study entry
* Previous use of an anti-VEGF drug in the study eye
* Cataract surgery or any other intraocular surgery in the study eye within 3 months prior to study entry
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 30 mm Hg despite treatment with maximal anti-glaucoma medications)
* History of stroke, myocardial infarction, transient ischemic attacks within 3 months prior to the study
* Pregnancy (positive urine pregnancy test) or lactation
* The presence of active malignancy, including lymphoproliferative disorders.
* History of allergy to fluorescein or any component of the ranibizumab formulation
* Active intraocular infection
* Participation in another simultaneous interventional medical investigation or trial
* Women with child bearing potency without effective contraception (i. e. implants, injectables, combined oral contraceptives, some IUDs or vasectomised partner) during the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint is the time to treatment success | up-to 29 months
  Time from randomisation until the date of last criteria-based intravitreal injection in case that thereafter a treatment-free period for (at least) 6 months was observed.

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | Month 29
  Best corrected visual acuity (BCVA) in number of ETDRS letters (Early Treatment of Diabetes Retinopathy Study) per visit
Central subfield thickness (CST) | Month 29
  Central subfield thickness (CST) measured by OCT per visit
Number of ranibizumab injections | Month 29
  Number of ranibizumab injections required until treatment success and up to the end of Observation.

OTHER OUTCOMES:
Development of neovascularization(s) | Month 24
  Proportion of subjects developing neovascularization(s) of retina, optic disc, and/or in anterior segment over the total period of observation.
The area of non-perfusion | Month 24
  The area of non-perfusion (assessed by FA) will be quantified as sum of all areas identified
Vessel density | Month 24
  Assessed by OCT-angiography, will be quantified by a metric measure with the range [0;1]
Potential visual field loss | Month 4 and Month 24
  The change between the two timepoints (Months 4 and 24) per arm will be used to characterize the both groups and be compared between treatment arms.
The number of laser treatments and the laser spots given in the experimental group (RL-arm). | Month 24
  The number of visits with applied laser treatment and the laser spots applied in the experimental group (RL-arm) will be counted for descriptive reasons and be compared between treatment arms.
Health-related quality of life (QoL): Visual Function Questionnaire VFQ25 | Baseline, Month 12 and Month 24
  Measured by the Visual Function Questionnaire VFQ25
Areal of foveal avascular zone | Month 24
  Area of the foveal avascular zone (FAZ, assessed by OCT-angiography, will be quantified in [mmm²])

CONTACTS AND LOCATIONS:
Overall Officials: Matus Rehak, Professor, Study Director — Department of Ophthalmology Justus-Liebig-Universität Giessen
Locations (15):
- Medizinische Universität Innsbruck, Klinik für Augenheilkunde und Optometrie, Innsbruck, Austria
- Germany (14):
  - Universitätsklinikum Carl Gustav Carus Dresden Klinik und Polyklinik für Augenheilkunde, Dresden
  - Internationale Innovative Ophthalmochirurgie GbR, Klinik für Augenchirurgie, Düsseldorf
  - Universitätsklinikum Klinik für Augenheilkunde Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen, Klinik und Poliklinik für Augenheilkunde, Giessen
  - Hannover MHH Universitätsklinik für Augenheilkunde, Hanover
  - University Hospital of Leipzig Department of Ophthalmology, Leipzig
  - Klinikum der Stadt Ludwigshafen Augenklinik, Ludwigshafen
  - Universitätsklinikum Gießen und Marburg GmbH, Standort Marburg Klinik für Augenheilkunde, Marburg
  - Ludwig-Maximilians-Universität München, Augenklinik, München
  - Augenzentrum am St. Franziskus-Hospital Münster, Münster
  - Universitätsklinikum Klinik für Augenheilkunde, Münster
  - Universitätsklinikum Tübingen, Department für Augenheilkunde, Tübingen
  - Universitätsklinikum Ulm, Klinik für Augenheilkunde, Ulm
  - Augen-OP-Zentrum Zschopau, Praxis für Augenheilkunde, Zschopau

DOCUMENTS (1):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT04444492/Prot_000.pdf